CLINICAL TRIAL: NCT04261634
Title: Comparison of Clinical Effects of Concentrated Growth Factor and Platelet-Rich Fibrin in the Treatment of Adjacent Multiple Gingival Recessions: A Split-Mouth Randomized Clinical Trial
Brief Title: CGF and PRF in the Gingival Recessions Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Seyma Bozkurt Doğan, Associate Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 36290600/39
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Gingival Recession
Keywords: multiple gingival recession; platelet rich fibrin; concentrate growth factor
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentrated growth Factor Membrane (Experimental): Autogenous platelet and leukocyte fibrin material was obtained from blood.
  Interventions: Procedure: Concentrated Growth Factor Membrane; Procedure: Platelet Rich Fibrin
- Platelet Rich Fibrin (Active Comparator): Autogenous platelet and leukocyte fibrin material was obtained from blood.
  Interventions: Procedure: Concentrated Growth Factor Membrane; Procedure: Platelet Rich Fibrin

INTERVENTIONS:
Procedure: Concentrated Growth Factor Membrane — Concentrated growth factor is produced by the centrifugation of venous blood and platelets are concentrated in a gel layer containing fibrin matrix
  Other Names: An agent of platelet concentrates
Procedure: Platelet Rich Fibrin — Platelet Rich Fibrinis produced by the centrifugation of venous blood and platelets are concentrated in a gel layer containing fibrin matrix
  Other Names: An agent of platelet concentrates

SUMMARY:
This study hypothesized that CGFs' placement together with CAF may enhance the healing of soft tissues better than use of PRF together with CAF. Therefore, the aim of this study was to determine the clinical effects of CGF in combination with CAF compared to the clinical effect of PRF in combination with CAF in the treatment of adjacent multiple GRs.

DETAILED DESCRIPTION:
The gingival margin, which should be in the cemento-enamel junction (CEJ), migrates to the apical with the effect of many facilitating and triggering etiological factors. As a result of gingival recessions (GRs), the root surface (RS) is exposed, root hypersensitivity, root caries and cervical abrasion may occur, plaque control become difficult, resulting in a non-aesthetic appearance. Platelet concentrates (PCs) increase wound healing and repair by mediating the release of growth factors (GFs), such as platelet-derived GF, fibroblast GF, transforming GF-beta and insulin-like GF-I. These GFs were released from the local application of PCs which may enable better tissue regeneration and repair in dental and medical area.

Platelet-Rich Fibrin (PRF) has a more elastic and more sturdy membrane structure, which is rich in platelets and leucocytes.Concentrated growth factor (CGF) is an another generation of PCs. It is produced by the centrifugation of venous blood and platelets are concentrated in a gel layer containing ﬁbrin matrix as same as PRF. This study hypothesized that CGFs' placement together with (coronally advanced flap) CAF may enhance the healing of soft tissues better than use of PRF together with CAF. Therefore, the aim of this study was to determine the clinical effects of CGF in combination with CAF compared to the clinical effect of PRF in combination with CAF in the treatment of adjacent multiple GRs.

The patients of this randomized, split-mouth and controlled clinical trial study protocol were selected from individuals referred to the Department of Periodontology, at the Faculty of Dentistry, Bulent Ecevit University, for either dentin hypersensitivity or aesthetic complaints between May 2015 and June 2016.

The subjects were enrolled to this study based on the following inclusion criteria: (1) age > 18 years, (2) systemically and periodontally healthy, (3) non-smokers, (4) presence of ≥2 buccal adjacent Miller Class I or II GR with ≥2 mm GR depth (RD), probing depth (PD) <3 mm and gingival thickness (GT) ≥1 mm on both sides of the maxillary arch, (5) width of keratinized gingiva (KGW) ≥2 mm, (6) presence of identiﬁable cemento-enamel junction CEJ, (7) central, lateral canine and premolar teeth with GRs in the maxilla (8) full-mouth plaque control record (PCR) ≤20% (O'Leary et al. 1972) and gingival index (GI) scores = 0 (Loe, 1967) and presence of tooth vitality and absence of caries, restorations and furcation involvement in the treated area.

All the subjects received oral hygiene instructions and full-mouth scaling were performed 1 month before surgery. They were instructed to perform a non-traumatic brushing technique (Roll) using an ultra-soft toothbrush. In eighteen patients (mean age 39.67₊10.25 age; 8 females, 10 males), one side of the jaw received PRF+ CAF (37 defects), the opposite site received CGF + CAF (39 defects).

Application of PRF membrane to the control region: The patient's venous blood was taken into the 10-ml test tubes and placed quickly in the Electro-Mag centrifuge (M 815 P, İstanbul, Turkey) without shaking. The device was operated at 2700 rpm for 12 minutes to obtain PRF. Application of CGF membrane to the test region: The intravenous blood of the patient was taken into 10-ml glaas-coated test tubes without anticoagulant solutions and rapidly centrifuged with a CGF centrifuge machine (Medifuge, Silfradent, S. Sofia, Italy). The instrument's CGF program was selected and operated at speeds and angles ranging from 2700 to 3000 rpm. After approximately 13 minutes of rotation, CGF was obtained. CGF is characterized by 4 phases: (1) serum in the top layer, (2) the second buffy coat layer, (3) the third GF and unipotent stem cell layer (CGF), (4) the lower red blood cell layer (RBC). The CGFand PRF clot was removed from the tube and separated from the RBC by using microsurgical scissors. The CGF was squeezed in a special box that produces membranes at a constant thickness of 1 mm.All surgeries were performed by the same expert periodontist during a single surgical session Gingival recession sites were randomly determined as either test or control site by tossing a coin immediately before the surgical procedure.

Sutures were removed after 10 days and plaque control was maintained by CHX for additional 2 weeks. The patients started brush the tooth at the end of the 3rd week and they were again instructed in mechanical tooth cleaning of the treated tooth using an ultra soft toothbrush and roll technique. Oral hygiene instructions were provided at each postoperative visit.

ELIGIBILITY:
Inclusion Criteria:

* systemically and periodontally healthy,
* non-smokers
* presence of ≥ 2 buccal adjacent Miller Class I and II gingival recession with ≥ 2 mm gingival recession depth , probing depth <3 mm and gingival thickness (GT) ≥ 1 mm on both sides of the maxillary arch
* width of keratinized gingiva ≥ 2mm
* presence of identifiable cemento-enamel junction
* full-mouth plaque index (PI) < 20 % and gingival index (GI) scores <1,
* presence of tooth vitality and absence of caries, restorations and furcation involvement in the treated area,

Exclusion Criteria:

* patients who had systemic problems that wound contraindicate for periodontal surgery, - usage of medications known to interfere with healing and to cause gingival enlargement - recession defects associated with demineralization, deep abrasion,
* previous surgery in the defects area within the past 1 year,
* pregnant or lactating females
* drug and alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Complete root coverage | 6 months
  Change from baseline in percentage of complete root coverage at 6th months.

SECONDARY OUTCOMES:
Percentage root coverage | 6 months
  Change from baseline in percentage of complete root coverage at 6th months.
Keratinized gingiva width | 6 months
  The distance is from the mucogingival junction (MGJ) to the gingival margin
Recession depth | 6 th months
  The distance is from the cemento-enamel junction to the gingival margin
Probing depth | 6 th months
  The distance is from the gingival margin to the bottom of the sulcus